CLINICAL TRIAL: NCT03293966
Title: Therapeutic CARE of the Bronchial Cancer Not in Small Cell: Security of the Dispensation of Medicine by the Implementation of a Card of Coordination of Care Relative to the Medicinal Treatments Got Out of it From Hospitalization
Brief Title: A Coordination Card of Care Relative to the Medicinal Treatments Got Out of it From Hospitalization
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRIMACIE
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Treatment Related Cancer
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The continuity of the medicinal care between the city and the hospital stays a major organizational stake and of safety of patients' therapeutic care.This takeover is more complex when it concerns pathology needed lots of hospitalization and included the intervention of multiple healthcare practionners. This is clearly the case of cancer coverage.

The optimization of the therapeutic suppor in town is based on pharmaceutical advice strengthening but also on the pharmaceutical analysis to check the entire treatments' prescription and eventual medicinal interactions which ensue from it.That's why it's important to have a medicinal conciliation that takes into account all the medecine taken or have to be taken by the patient.

A specific support was developped by nurses , doctors and pharmacist ; it's a care coordination card that can be put easely in a pocket by the patient.

The aim of the study is that this card can be also used as a communication tools by sharing the prescription done at the release of hospital by using an IT link (flea datamatrix) for the patients Via the use of an IT link (flea datamatrix) for the patients whose pathology is complex in term of extra hospital coverage.

DETAILED DESCRIPTION:
The aim of this strudy is to evaluate with community pharmacists the impact of a new information system on the prevalence of dispensing difficulties reported by pharmacies when hospitalized patients leave the city. This information system will be based on the care coordination card implemented by a secure computer link allowing the use of information on treatments prescribed at the end of hospitalization. Patient management is not changed by this protocol. Only the information of the pharmacist, which is the object of the study, is increased.

ELIGIBILITY:
Inclusion Criteria:

* all patient admitted in onco-thoracic service
* Handled by an anticancer agent
* Having frequented the same city pharmacy for at least 3 months

Exclusion Criteria:

* hospitalization above 21 days
* refusing participation
* palliative care
* misunderstanding of french language
* frequenting several pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to thoracic pneumology and oncology treated with anticancer drugs will receive a medication conciliation.
  Patients integrating the study will be patients who have benefited from the entire process of medication conciliation (entry and exit) and returning home.
  The included patients must have attended the same pharmacy for at least 3 months (according to the patient declaration).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Composite criteria including all the dysfunctions noticed at the release of the hospital prescription intended to be dispensed in town. | 7days+/- 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France